CLINICAL TRIAL: NCT07235618
Title: A Phase II, Two-Stage Study Evaluating the Efficacy of Entinostat in Combined With Fulvestrant in Locally Advanced or Metastatic Breast Cancer With Recurrence or Progression After CDK4/6 Inhibitor Plus Endocrine Therapy
Brief Title: A Study of Entinostat in Combination With Fulvestrant for the Treatment of Locally Advanced or Metastatic Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, wang shusen, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EOC103D201
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced or Metastatic Breast Cancer
Keywords: Locally Advanced or Metastatic Breast Cancer; Entinostat; Fulvestrant; HR positive and HER2 negtive
MeSH Terms: conditions — Breast Neoplasms | interventions — entinostat; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Entinostat + Fulvestrant (Experimental)
  Interventions: Drug: Entinostat; Drug: Fulvestrant

INTERVENTIONS:
Drug: Entinostat — Entinostat (5mg/week, po)
Drug: Fulvestrant — Fulvestrant( 500 mg intramuscularly on Days 1 and 15 of Cycle 1, and then on Day 1 of each subsequent 28-day cycle)

SUMMARY:
This study aims to evaluate the efficacy of Entinostat combined with Fulvestrant in HR+/HER2- advanced breast cancer patients with recurrence/progression after endocrine therapy (primary endpoint: progression-free survival [PFS]), and explore the correlation between peripheral blood mononuclear cell (PBMC) acetylation levels and treatment response to determine the baseline acetylation threshold .

ELIGIBILITY:
Inclusion criteria：

1. Signed informed consent form.
2. Female participants aged ≥18 and ≤75 years. 3 .Eastern Cooperative Oncology Group (ECOG) performance status of 0-1

4. Life expectancy ≥3 months. 5.Participants must have histopathologically and molecular pathologically diagnosised HR-positive and HER2-negative breast cancer (based on the most recent report),defined as presence of following criteria:

1. . Hormone receptor positivity is defined by the presence of estrogen receptors (ER), where a threshold of ≥10% positive staining cells is considered indicative of positivity. The status of progesterone receptors (PR) can be either negative or positive, with the same criterion of ≥10% positive staining cells applied to determine receptor positivity.
2. . HER-2 negativity indicates that the immunohistochemical assessment of the pathological specimen yields a result classified as 0 or 1+. Alternatively, a result classified as 2+ may also be deemed HER-2 negative if corroborated by negative findings from ISH or FISH testing.

6. Participants must have received endocrine +CDK4/6 inhibitor treatment and meet any of the following conditions, namely endocrine resistance:

a) Imaging progression occurs during adjuvant/neoadjuvant endocrine therapy; or b) Recurrence/metastasis within ≤12 months after the completion of adjuvant endocrine therapy; or c) Disease progression occurred after first-line endocrine therapy in the advanced stage (RECIST v1.1).

7.Prior chemotherapy history for the participants must meet:

1. For metastatic diseases, having received ≤1 line of chemotherapy (including antibody-drug conjugates) in the past;
2. The period from the end of the last chemotherapy administration to the randomization date is ≥4 weeks;
3. If disease progression occurs within ≤12 months after the end of neoadjuvant or adjuvant chemotherapy, this regimen is regarded as first-line chemotherapy in the metastasis stage.

   8.One week (7 days) before the start of the study administration, the participant must have adequate organ function, as defined below: Hematology: Hemoglobin (HgB) ≥80 g/L, platelet count ≥50×109 /L, absolute neutrophil count ≥1.0×109 /L.

   Note: Before these laboratory tests, platelet transfusion is not allowed within 3 days, red blood cell transfusion is not allowed within 14 days, and hematopoietic growth factor (pegylated G-CSF and erythropoietin within 14 days) is not allowed within 7 days.

   Renal function: Serum creatinine (Cre) ≤1.5× upper limit of normal (ULN), or glomerular filtration rate (eGFR) ≥60 mL/min/1.73m2.

   Liver function: Total bilirubin ≤1.5×ULN; If Gilbert syndrome is present, the total bilirubin is ≤3 mg/dL. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3×ULN; If there is liver metastasis, both ALT and AST should be ≤5×ULN. Alkaline phosphatase (ALP) ≤2.5×ULN; If there is bone metastasis, it should be ≤5×ULN.

   9.Left ventricular ejection fraction (LVEF) ≥50% by echocardiogram and QTc interval ≤480 ms.

   10.Female participants in the premenopausal or perimenopausal stages who consent to the use of concomitant luteinizing hormone-releasing hormone (LHRH) agonists are eligible for enrollment. Participants meeting any of the following criteria may be classified as having reached menopause; those not fulfilling these criteria will be considered to be in the premenopausal or perimenopausal period:

   1)- A history of bilateral oophorectomy; 2）- Age ≥ 60 years; 3）- Age < 60 years, with natural amenorrhea lasting ≥ 12 months, during which no chemotherapy, tamoxifen, torremifene, or ovarian castration was administered. Additionally, blood levels of follicle-stimulating hormone (FSH) and estradiol (E2) must fall within the postmenopausal range (as determined in conjunction with the reference range established by the research center); 11.Participants of childbearing potential must use effective contraception (e.g., spermicidal condoms, vaginal diaphragm, oral/injectable contraceptives) or practice abstinence during and for 3 months after treatment.

   Exclusion criteria：
   1. Presence of current or prior Central Nervous System (CNS) metastases or leptomeningeal disease (LMD).
   2. Prior treatment with Selective Estrogen Receptor Degraders (SERD, e.g., fulvestrant) or Histone Deacetylase (HDAC) inhibitors (e.g., entinostat, chidamide).
   3. Known to be allergic to SERD, entinostat or other drugs with a benzamide structure (such as tyapride, remopilib, cloprapride, etc.).
   4. Pregnant or lactating women.
   5. Combined with other malignant tumors, unless radical treatment has been carried out and there is no evidence of recurrence or metastasis;
   6. Clinically significant effusions requiring drainage (e.g., pericardial, pleural, or ascites with symptoms).
   7. Significant clinical gastrointestinal dysfunction that may affect oral medication intake, transport, or absorption(e.g., dysphagia, chronic diarrhea, intestinal obstruction).
   8. Severe infectious diseases, uncontrolled or severe cardiovascular diseases, or other abnormalities within 14 days before enrollment that the investigators considered might affect the safety and compliance of the subjects and were not suitable for participation in this clinical trial.
   9. Participants deemed by investigators as unsuitable for endocrine therapy.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to 1 year
  Progression-free survival(PFS) is defined as the time from treatment initiation to disease progression or death from any cause.

SECONDARY OUTCOMES:
Overall Survival(OS) | Up to 3 years
  Overall survival (OS) is defined as the time from treatment initiation to death from any cause.
Objective Response Rate(ORR) | Up to 3 years
  Objective response rate (ORR) is defined as the percetage of participants achieving a complete response (CR) or partial response (PR) according to RECIST v.1.1.
Clinical Benefit Rate(CBR) | Up to 3 years
  Clinical Benefit Rate(CBR) is defined as the percetage of participants achieving a complete response (CR) and partial response (PR) and stable disease （SD）≥ 24 weeks according to RECIST v.1.1.
Duration of response(DOR) | Up to 3 years
  Duration of response (DOR) is defined as the duration from response initiation (when either CR or PR ) to progression or death, whichever occurs first.
Health-Related Quality of Life | Up to 3 years
  Quality of life measures will be assessed at baseline, the 28th day of the first cycle the 28th day of the fourth cycle, and the 28th day of each subsequent cycle, at the end of the treatment and will be collected using patient reported outcome questionnaires: Cancer Treatment Function Evaluation System - Breast Cancer (FACT-B)
Treatment compliance | Up to 3 years
  The proportion of high, medium and low adherence to each drug will be calculated along with the binomial exact 95% confidence interval.
Number of participants with adverse events | Up to 3 years
  Adverse events are assessed by CTCAE v5.0

OTHER OUTCOMES:
Biomarker analysis(protein lysine acetylation of peripheral blood samples (PBMCs)) | Up to 1 year
  Protein lysine acetylation of peripheral blood samples (PBMCs) will be assessed at baseline, the first day of the first cycle,the 15th day of the first cycle, the first day of the fourth cycle, and the 15th day of fourth cycle, at the end of the treatmentthe fourth cycle, and the 15th day of fourth cycle, at the end of the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No